CLINICAL TRIAL: NCT01279200
Title: Use of High Cost Monitoring During Letrozole Ovulation Induction and Effect on Pregnancy Rates - A Pilot Study
Brief Title: Use of High Cost Monitoring During Letrozole Ovulation Induction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Blue Cross Blue Shield of Michigan Foundation (Other)
Responsible Party: Principal Investigator, Senait Fisseha, MD, JD, Medical Director, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00041349; 1726.PIRAP (Other Grant/Funding Number: Blue Cross Blue Shield of Michigan Foundation)
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Results first posted 2015-01-06 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Infertility
Keywords: letrozole; ovulation monitoring; pregnancy rate
MeSH Terms: conditions — Infertility | interventions — Ovidrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Urinary LH Kits (Active Comparator): Patients randomized to this arm will monitor ovulation with home-based urinary LH kits (Ovulation Predictor Kits, OPK's).
  Interventions: Other: Urinary LH kits
- Midcycle ultrasound + hCG injection (Active Comparator): Patients randomized to this arm will undergo ovulation monitoring with midcycle ultrasound and receive hCG injection if evidence of a mature size follicle.
  Interventions: Other: Midcycle ultrasound + hCG injection

INTERVENTIONS:
Other: Midcycle ultrasound + hCG injection — Mid-cycle ultrasound with administration of hCG (single dose of standardized pre-filled injection, 250 mcg, at time of ultrasound) when appropriate.
  Other Names: Ovidrel
  Arms: Midcycle ultrasound + hCG injection
Other: Urinary LH kits — Subjects randomized to monitoring with LH kits at home will keep a monthly calendar documenting when LH testing begins, day LH surge occurs and day(s) of intercourse/insemination.
  Other Names: ClearBlue Easy
  Arms: Urinary LH Kits

SUMMARY:
The purpose of this study is to investigate monitoring methods during ovulation induction cycles with letrozole and their effect on pregnancy rates. Monitoring ovulation induction cycles with letrozole can be done with a variety of methods, the two most commonly utilized are home-based urinary LH kits (or ovulation predictor kits) and office-based midcycle follicular ultrasound. Letrozole coupled with follicular monitoring by ultrasound may add extra cost per cycle with no improvement in fecundability (pregnancy rates per cycle).

DETAILED DESCRIPTION:
The study will be a randomized controlled trial of adult women with primary and secondary infertility seen at the University of Michigan Health System undergoing ovulation induction (OI) with letrozole as part of their standard clinical care. Patients who are undergoing OI with letrozole as per standard clinical care will be randomized to urinary luteinizing hormone (LH) ovulation predictor kit use versus mid-cycle ultrasound with administration of hCG when appropriate for timing of intercourse or intrauterine insemination. Patients who have been prescribed letrozole as per routine clinical care will be approached to determine willingness to participate in this study. Study period involves up to three ovulation induction cycles or until pregnancy occurs.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 21-39 undergoing letrozole ovulation induction (as part of routine clinical care) at a single academic-infertility center.
* Normal uterus and evidence of at least tubal patency on one side (as assessed by saline-infusion sonography or hysterosalpingogram per clinical care).

Exclusion Criteria:

* Current pregnancy
* Nursing mothers
* Prior hypersensitivity to hCG preparations
* Primary ovarian failure or menopausal levels of FSH (>12 mIU/mL)
* Patients with abnormal uterine bleeding of undetermined origin or ovarian cyst of undetermined origin, sex-hormone dependent tumors, documented bilateral tubal obstruction, uncorrected uterine anomalies,
* Previous letrozole or gonadotropin use and/or previous treatment with in vitro fertilization
* Other uncorrected medical condition that would be a contraindication to attempting elective ovulation induction (e.g., uncontrolled diabetes, intracranial lesion, thyroid or adrenal disease).

Ages: 21 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2011-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senait Fisseha, MD, JD, Principal Investigator — University of Michigan
Locations (1):
- Center for Reproductive Medicine, University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Pritts EA. Letrozole for ovulation induction and controlled ovarian hyperstimulation. Curr Opin Obstet Gynecol. 2010 Aug;22(4):289-94. doi: 10.1097/GCO.0b013e32833beebf. PMID 20592587
- [Background] Mitwally MF, Casper RF. Use of an aromatase inhibitor for induction of ovulation in patients with an inadequate response to clomiphene citrate. Fertil Steril. 2001 Feb;75(2):305-9. doi: 10.1016/s0015-0282(00)01705-2. PMID 11172831
- [Background] Mitwally MF, Abdel-Razeq S, Casper RF. Human chorionic gonadotropin administration is associated with high pregnancy rates during ovarian stimulation and timed intercourse or intrauterine insemination. Reprod Biol Endocrinol. 2004 Jul 7;2:55. doi: 10.1186/1477-7827-2-55. PMID 15239837
- [Background] Deaton JL, Clark RR, Pittaway DE, Herbst P, Bauguess P. Clomiphene citrate ovulation induction in combination with a timed intrauterine insemination: the value of urinary luteinizing hormone versus human chorionic gonadotropin timing. Fertil Steril. 1997 Jul;68(1):43-7. doi: 10.1016/s0015-0282(97)81473-2. PMID 9207582
- [Background] Zreik TG, Garcia-Velasco JA, Habboosh MS, Olive DL, Arici A. Prospective, randomized, crossover study to evaluate the benefit of human chorionic gonadotropin-timed versus urinary luteinizing hormone-timed intrauterine inseminations in clomiphene citrate-stimulated treatment cycles. Fertil Steril. 1999 Jun;71(6):1070-4. doi: 10.1016/s0015-0282(99)00116-8. PMID 10360912
- [Background] Lewis V, Queenan J Jr, Hoeger K, Stevens J, Guzick DS. Clomiphene citrate monitoring for intrauterine insemination timing: a randomized trial. Fertil Steril. 2006 Feb;85(2):401-6. doi: 10.1016/j.fertnstert.2005.07.1331. PMID 16595218
- [Background] Smith YR, Randolph JF Jr, Christman GM, Ansbacher R, Howe DM, Hurd WW. Comparison of low-technology and high-technology monitoring of clomiphene citrate ovulation induction. Fertil Steril. 1998 Jul;70(1):165-8. doi: 10.1016/s0015-0282(98)00119-8. PMID 9660442

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Urinary LH Kits | Midcycle Ultrasound + hCG Injection
Started | 10 | 11
Completed | 8 | 4
Not Completed | 2 | 7
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Patient withdrawal due to high cost | 0 | 1
Not completed — Inconvenience of ultrasound visit | 0 | 1
Not completed — ultrasound screening failure | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Urinary LH Kits | Midcycle Ultrasound + hCG Injection | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Mean (Full Range); unit: years] | 28.7 [21 to 39] | 29.8 [21 to 39] | 29.3 [21 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 9 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Gravidity: number of previous pregnancies [Mean (Full Range); unit: pregnancies] | .7 [0 to 2] | 1.1 [0 to 4] | .9 [0 to 4]
Diagnosis of ovulatory dysfunction [Number; unit: participants]
  prior diagnosis of ovulatory dysfunction | 4 | 3 | 7
  no prior diagnosis of ovulatory dysfunction | 6 | 8 | 14

OUTCOME MEASURES:

1. Secondary Outcome: Time to Conception, Measured in Cycles
Description: Cycles means treatment/menstrual cycles, approximately 28-33 days.
Time Frame: 3 menstrual/treatment cycles, or upon conception, whichever comes first
Population: Numbers of participants analyzed changes from 8 with kits and 4 with ultrasound (enrolled) because time to conception can be measured only for those who conceived, so the 6 and 1 participants analyzed here are those who were successful in getting pregnant.
Measure: Mean (Full Range); unit: menstrual cycles
Arm/Group | Urinary LH Kits | Midcycle Ultrasound + hCG Injection
Number analyzed (Participants) | 6 | 1
menstrual cycles | 1.83 [1 to 3] | 1 [1 to 1]

2. Primary Outcome: Pregnancy Success Rate
Description: Percentage of women in each arm who became pregnant within the study time frame.
Time Frame: 3 menstrual/treatment cycles (approximately 28-33 days each)
Measure: Number; unit: percentage of participants
Arm/Group | Urinary LH Kits | Midcycle Ultrasound + hCG Injection
Number analyzed (Participants) | 8 | 4
percentage of participants | 75 | 25

ADVERSE EVENTS:
Time Frame: End of Cycle 1, Cycle 2 and Cycle 3; OB ultrasound (if applicable); and at the End of Study visit.
Description: Phone call (group A) or in-person assessment (group B).
Arm/Group | Urinary LH Kits | Midcycle Ultrasound + hCG Injection
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 1/10 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Urinary LH Kits (N=10) | Midcycle Ultrasound + hCG Injection (N=11)
Side effects (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — bone pain, arthralgia

LIMITATIONS AND CAVEATS:
The original intent was to study 400 women, but due to recruiting and time restraints, final enrollment was only 21. Therefore, statistical analyses of the results were eliminated, as well as some additional outcome measures originally planned for.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes